CLINICAL TRIAL: NCT05777902
Title: Multidimensional Integrated Assessment of Neurological and Immunological Patterns to Test the Efficacy and Response to Ozanimod in Multiple Sclerosis.
Brief Title: Multidimensional Integrated Assessment to Test the Efficacy and Response to Ozanimod in Multiple Sclerosis.
Acronym: OMNIAOMS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EUDRACT 2021-005860-24
Record Dates: First submitted 2023-03-09; First posted 2023-03-21 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2023-02

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — ozanimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient (Experimental)
  Interventions: Drug: Ozanimod Oral Capsule

INTERVENTIONS:
Drug: Ozanimod Oral Capsule — We propose to integrate measurements obtained using multiple tools. Patients will undergo MRI and hdEEG procedures, and blood samples will be obtained for the immunological and biochemical studies on the same day. The study of the immune system's status will include an extensive immunophenotypic analysis, a functional characterization following ex vivo stimulation of innate immune cells, and the measurement of soluble products in the serum, such as cytokines. Cellular traits of interest include the absolute numbers and relative proportions of specific cell subsets, transcriptional states, secretory functions, proliferative capacity or cytolytic potential. Specifically, the following antibody combination will constitute the core of the immunophenotypic analysis: HLADR CD11c, CD38, CD14, CD123, lineage (CD3, CD56, CD19).
  Other Names: Zeposia

SUMMARY:
This is a prospective interventional study with a 12-month follow-up of patients diagnosed with Multiple Sclerosis. Enrollment includes patients for whom Ozanimod will be prescribed based on regular clinical practice. It is proposed to integrate the measurements obtained using multiple instruments, with the aim of analyzing the immunological landscape, connectivity networks and anatomical traits of neurodegeneration.

Patients will return for imaging and noninvasive electrophysiological studies 3, 6, and 12 months after initiation of therapy. On the same day, blood samples will be taken and immunological and biochemical tests will be performed.

DETAILED DESCRIPTION:
This is a prospective interventional study with a 12-month follow-up of patients diagnosed with Multiple Sclerosis. Enrollment includes patients for whom Ozanimod will be prescribed based on regular clinical practice. It is proposed to integrate the measurements obtained using multiple instruments, with the aim of analyzing the immunological landscape, connectivity networks and anatomical traits of neurodegeneration.

Patients will return for imaging and noninvasive electrophysiological studies 3, 6, and 12 months after initiation of therapy. On the same day, blood samples will be taken and immunological and biochemical tests will be performed.

The primary objective of the study is to use this multidimensional integrated approach to verify the therapeutical activity of Ozanimod on the inflammatory mediated neurodegeneration.

The endpoint that relate to this objective is to evaluate the innate immune mediated inflammation in MS patients and to correlate it with the cognitive reserve and with serum NFL levels before and after Ozanimod treatment.

Patients must meet all the following inclusion criteria to be eligible for enrolment into the study:

1. Diagnosis of MS accordingly to 2017 revised McDonald criteria;
2. Patients candidate to receive Ozanimod therapy (disease characteristics, EDSS, age, lifestyle, disease progression, etc.);
3. Age between 18 and 45 years;
4. EDSS score from 0 to 4;
5. Signature and date of written ICF prior to entering the study;

ELIGIBILITY:
Inclusion Criteria:

* 1) Diagnosis of MS accordingly to 2017 revised McDonald criteria; 2) Patients candidate to receive Ozanimod therapy (disease characteristics, EDSS, age, lifestyle, disease progression, etc.); 3) Age between 18 and 45 years; 4) EDSS score from 0 to 4; 5) Signature and date of written ICF prior to entering the study;

Exclusion Criteria:

* The presence of any of the following will exclude a patient from study enrolment:

  1. Ongoing immunomodulatory or immunosuppressive treatment;
  2. Other autoimmune comorbidities (i.e. antiphospolipid syndrome);
  3. Treatment with steroids in the last 30 days before enrollment;
  4. Acute inflammatory status not MS related (i.e. bacterial or viral infections) in the previous 30 days;
  5. Patients unable to read and understand the documents of the study.
  6. Participation in any interventional clinical trials or compassionate use programs
  7. Contraindications and "not-recommendations" reported in SmP

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-04-11 (Actual)

PRIMARY OUTCOMES:
verify the therapeutical activity of Ozanimod on the inflammatory mediated neurodegeneration. | 12 months
  To evaluate the innate immune mediated inflammation in MS patients and to correlate it with the cognitive reserve and with serum NFL levels before and afterOzanimod treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione Santa Lucia, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No